CLINICAL TRIAL: NCT06502561
Title: A Phase 1 Relative Bioavailability Study Comparing The Pharmacokinetics Of Aramchol Meglumine Granules For Oral Suspension To Aramchol Free Acid 300 mg Tablets In Healthy Volunteers
Brief Title: Comparing The PK Of Aramchol Meglumine Granules To Aramchol Free Acid Tablets
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AM-001
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Salts

STUDY DESIGN:
Intervention Model Description: All subjects will receive a single dose of 400 mg Aramchol meglumine granules for oral suspension (Test 1) in Period 1.
  In Periods 2 and 3, subjects will be randomized to a crossover of treatments in a 1:1 ratio to receive a single dose of Aramchol meglumine granules for oral suspension (Test 2) in one period and a 300 mg Aramchol free acid tablet (Reference) in the other period. The washout interval between dosing periods will be at least 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Subjects receiving a single 400 mg dose of Aramchol meglumine in Period 1 (Experimental): A single 400 mg dose of Aramchol meglumine will be administered to all study subjects in Period 1.
  Interventions: Drug: Aramchol meglumine
- Subjects receiving a second dose of Aramchol meglumine or Aramchol free acid in Period 2 (Active Comparator): In Period 2, study subjects will be randomized 1:1 to receive Aramchol meglumine or 300 mg tablet of Aramchol free acid (Reference)
  Interventions: Drug: Aramchol meglumine; Drug: Aramchol free acid
- Subjects receiving a second dose of Aramchol meglumine or Aramchol free acid in Period 3 (Active Comparator): In Period 3, study subjects will be randomized 1:1 to receive Aramchol meglumine or 300 mg tablet of Aramchol free acid (Reference)
  Interventions: Drug: Aramchol meglumine; Drug: Aramchol free acid

INTERVENTIONS:
Drug: Aramchol meglumine — Aramchol meglumine is a salt form of Aramchol free acid
  Other Names: Cholan-24-oic acid 7,12-dihydroxy3-[(1-oxoeicosyl)amino]-(3β,5β,7α,12α) salt with N-methyl-(D)-glucamine-Aramchol Meglumine
Drug: Aramchol free acid — Aramchol free acid is a fatty acid-bile acid conjugate
  Other Names: 3β-arachidylamido-7α,12α-dihydroxy-5β-cholan-24-oic acid
  Arms: Subjects receiving a second dose of Aramchol meglumine or Aramchol free acid in Period 2; Subjects receiving a second dose of Aramchol meglumine or Aramchol free acid in Period 3

SUMMARY:
This is a Phase 1 Relative Bioavailability Study Comparing The Pharmacokinetics Of Aramchol Meglumine Granules For Oral Suspension To Aramchol Free Acid 300 mg Tablets In Healthy Volunteers

DETAILED DESCRIPTION:
A single center, 3-period, open-label, crossover study in healthy male and female volunteers who will receive 2 single doses of Aramchol meglumine and 1 single dose of Aramchol free acid under fasting conditions. A single 400 mg dose of Aramchol meglumine (Test 1) will be administered to all study subjects in Period 1. The second dose of Aramchol meglumine will be between 200 mg and 800 mg and will be selected after review of the pharmacokinetics (PK) from Period 1. In Periods 2 and 3, study subjects will be randomized 1:1 to receive the second dose of Aramchol meglumine (Test 2) in one period and a 300 mg tablet of Aramchol free acid (Reference) in the other period. Each product will be given under fasting conditions. The study periods will be separated by a wash-out period of at least 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects
2. Age between 18 and 45 years (inclusive of the date of signing the informed consent form)
3. Male subjects must be using two acceptable methods of contraception (e.g., spermicidal gel plus condom) for the entire duration of the study, and up to the study completion visit
4. Female subjects who are not of reproductive potential. A female subject who is not of reproductive potential is defined as a subject who:

   (i) has reached natural menopause (defined as at least 12 months of spontaneous amenorrhea); (ii) is at least 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy; or (iii) has undergone bilateral tubal ligation. Spontaneous amenorrhea does not include cases for which there is an underlying cause (e.g., anorexia nervosa).
5. Female subjects who are of reproductive potential and use reliable contraception method and/or are willing to use adequate birth control methods starting from at least 4 weeks prior to the screening visit and for the duration of the study through 30 days after the last dose of study drug

   List of medically accepted contraceptive methods:
   * Combination of a barrier method and spermicides (film, jelly, foam): female/ male condoms with spermicides, as well as a diaphragm/ cervical cap/ contraceptive sponge with spermicides.
   * Hormonal methods: combined estrogen/progestin injectable and oral contraceptives; progestin injectable and oral contraceptives; implants (Nexplanon®), vaginal ring (NuvaRing®), skin patch (Xulane®) and contraceptive injection (Depo-Provera®).
   * Intrauterine devices (IUD): inert or copper IUD (ParaGard®), hormonal IUD (Mirena®, Skyla®, Kyleena®).
6. Physically and mentally healthy as judged by means of medical and standard laboratory examinations
7. Non-smokers or ex-smokers (stopped at least 12 months ago) and non-users of other nicotine containing products, confirmed by urine cotinine test
8. Body mass index (BMI) within the range (including the borders) of 18.0 to 29.9 kg/m2
9. Informed consent given in written form according to Section 5.3 of clinical study protocol

Exclusion Criteria:

1. Participation in another clinical study at the same time or within 90 days before the screening visit (calculated from the date of the final examination of the previous study)
2. Randomization into the present study more than once
3. Blood donation or blood loss including plasmapheresis of >500 mL within 90 days before screening visit
4. History of drug abuse or use of illegal drugs: use of soft drugs, marihuana within 6 months before screening visit or hard drugs, cocaine, amphetamines, phencyclidine within 1 year before screening visit
5. Alcohol abuse, regular use of more than 2 units of alcohol per day or 10 units per week or a history of alcoholism (one unit of alcohol equals 250 mL beer, 125 mL wine or 25 mL spirits) or recovered alcoholics
6. Regular consumption of beverages or food containing methylxanthines (coffee, tea, cola, caffeine containing sodas, chocolate) equivalent to more than 500 mg methylxanthines per day
7. Positive drug screen
8. Positive alcohol test
9. Pregnant and/or nursing women. Positive pregnancy hCG test
10. Allergic diathesis or any clinically significant allergic disease (asthma or bronchial hyperreactivity)
11. Any history of drug hypersensitivity especially to the active and inactive ingredients of the Aramchol meglumine or Aramchol free acid preparations, including cholic acid
12. Presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, hematological, gastrointestinal, neurological, psychiatric or other diseases
13. Clinically significant illness within 4 weeks before screening visit
14. Major surgery of the gastrointestinal tract except for appendectomy
15. Any chronic disease which might interfere with absorption, distribution, metabolism or excretion of the drug
16. History of difficulty in swallowing
17. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies
18. Administration of depot injectable solutions or medications with a half-life > 1 week (including study medications) within 3 months before screening visit
19. Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before screening visit
20. Intake or administration of any oral, systemic or topical medication (including Over The Counter - OTC medication other than paracetamol and especially intake of antacids: aluminum hydroxide, magnesium hydroxide, and simethicone or herbal medication: St. John's wort, kava kava) within 2 weeks before screening visit
21. Vaccination within 14 days prior to screening visit
22. Medication with drugs known to alter the major organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within 60 days before screening visit
23. Systolic blood pressure outside the range of 100 to 140 mmHg and/or diastolic blood pressure outside the range of 60 to 90 mmHg
24. Pulse rate outside the range of 45 to 100 beats/min
25. Axillary body temperature outside the interval of 35.5 to 37.0°C
26. Any clinically significant abnormality of the resting 12-lead Electrocardiogram (ECG)
27. Laboratory values outside the normal range with clinical relevance
28. Special diet due to any reason (vegetarian)
29. Body weight loss of more than 10 kg in the last two months
30. History or presence of piercings in the mouth (tongue, lips) or wearing braces or dentures
31. Subjects who are known or suspected:

    * not to comply with the study directives
    * not to be reliable or trustworthy
    * not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed
    * to be in such a precarious financial situation that they no longer are able to weigh up the possible risks of their participation and the unpleasantness they may be involved in
    * subject is in custody or submitted to an institution due to a judicial order.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cmax of Aramchol | 10 weeks
  Observed maximal concentration after administration
AUClast of Aramchol | 10 weeks
  Area under the concentration/time curve, calculated by the trapezoidal rule from time 0 h to last observed concentration at time t
AUCinf of Aramchol | 10 weeks
  Area under the concentration/time curve, from time 0 h extrapolated to infinity

SECONDARY OUTCOMES:
Tmax of Aramchol | 10 weeks
  Observed time point of maximal concentration
λz of Aramchol | 10 weeks
  Terminal rate constant
t½ of Aramchol | 10 weeks
  Plasma concentration half-life
CL/F of Aramchol | 10 weeks
  Clearance per fraction of bioavailability
VZ/F of Aramchol | 10 weeks
  Volume of distribution per fraction of bioavailability
%AUCextrap of Aramchol | 10 weeks
  The percentage of the area under the concentration-time curve (%AUC) that is extrapolated beyond the last observed data point

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Gliut, MD, Principal Investigator — Project management
Locations (1):
- Diagnostic & Consultative Centre 'Ascendent' Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No